Official Title: The Impact of Cigarillo Warnings on Purchasing Behaviors Among Young Adult Cigarillo Users NCT05434013

IRB-Approved Date:4/7/2022

## Online Tobacco Marketplace Study Informed Consent to Participate in Research Jennifer Cornacchione Ross, PhD, Principal Investigator

You are invited to complete a survey as part of a research study being conducted by Wake Forest School of Medicine. The goal of the survey is to understand what young adults think about some tobacco products. You will complete a series of hypothetical purchasing tasks within a virtual online shopping marketplace. The survey will take about 15-20 minutes to complete.

We expect about 1,575 people to complete the survey. There is no cost to take the survey. After you complete the survey, you will earn approximately 100 Kantar points.

Taking part in this study is voluntary. You may choose not to take part or you may leave the study at any time. Refusing to participate in the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff. You will be given any new information we become aware of that would affect your willingness to continue to participate in the study.

There is minimal risk to you for completing the survey. You are not expected to personally benefit from this survey, but the results may help others in the future.

In this research study, any new information we collect from you about your health or behaviors is considered Protected Health Information. The information we collect for this research study includes age, state of residence, and tobacco use. We will make every effort to keep your Protected Health Information private. We will store records of your Protected Health Information on a password protected computer. Your Protected Health Information will not be shared outside our study team.

We will not collect any identifying information, such as your name, in this survey. Your participation is completely voluntary. You may stop taking the survey at any time. Your answers to this survey are completely confidential and will NOT be shared with anyone. Confidentiality will be protected by maintaining all study information in a secure manner. Data access will be limited to study staff. Data and records will be kept locked and secured, with any electronic data password protected. If you do not want to answer a question, you may skip it. No reference to any individual participant will appear in reports, presentations, or publications that may arise from the study.

If you have any questions, suggestions, or concerns regarding this survey, or if you wish to withdraw from the study, please contact the Principal Investigator Jennifer Cornacchione Ross at jcornacc@wakehealth.edu. If you have any questions, suggestions, or concerns regarding your rights as a participant in this study, please contact the Institutional Review Board at Forest at

By selecting "I Agree":

- You have read the above information
- You voluntarily agree to participate
- You are at least 18 years of age

Select "I Agree" if you would like to participate:

o I Agree